CLINICAL TRIAL: NCT00687219
Title: Treatment of Patients With Compensated Liver Cirrhosis With SCH 54031 + Ribavirin
Brief Title: Efficacy and Safety of Peginterferon Alfa-2b and Ribavirin Therapy in Subjects With Type C Compensated Liver Cirrhosis (Study P05116)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P05116; JPC-06-320-35
Record Dates: First submitted 2008-05-27; First posted 2008-05-30 (Estimated); Results first posted 2011-12-02 (Estimated); Last update posted 2017-04-07 (Actual); Status verified 2017-03

CONDITIONS: Hepatitis C, Chronic; Liver Cirrhosis
Keywords: hepatitis C
MeSH Terms: conditions — Hepatitis C, Chronic; Liver Cirrhosis; Hepatitis C | interventions — peginterferon alfa-2b; Ribavirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Peginterferon alfa-2b + Ribavirin (Experimental)
  Interventions: Biological: Peginterferon alfa-2b; Drug: Ribavirin

INTERVENTIONS:
Biological: Peginterferon alfa-2b — Administered at 1.0 µg/kg/week SC for 48 weeks
  Other Names: SCH 054031
Drug: Ribavirin — Administered based on body weight and hemoglobin value at Screening: 600-1000 mg/day for subjects with hemoglobin value at screening >=14g/dL, and 400-800 mg/day for subjects with hemoglobin value at screening >=12g/dL and <14g/dL; treatment duration is 48 weeks
  Other Names: SCH 018908

SUMMARY:
The objective is to evaluate the efficacy and safety of combination therapy with peginterferon alfa-2b 1.0 µg/kg/week subcutaneous (SC) + ribavirin administered for 48 weeks in participants with chronic hepatitis C and type C compensated liver cirrhosis. Participants who are hepatitis C virus ribonucleic acid (HCV-RNA) positive after 24 weeks of treatment will be discontinued from therapy.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 20-70 years.
* Positive quantitative serum HCV-RNA.
* Participants classified as A in Child-Pugh classification, and who do not have ascites or hepatic encephalopathy.
* Diagnosed with type C compensated liver cirrhosis based on liver biopsy performed within 3 years or latest celioscopy.
* Prolonged prothrombin time by <=3.0 sec.
* Participants and partners of participants willing to use adequate contraception during the course of the study.
* Participants who can be hospitalized for at least 14 days since treatment initiation.
* Weight >40 kg and <=100 kg
* Hematology laboratory results of:

  * hemoglobin >=12 g/dL
  * neutrophil count >=1,500/mm^3
  * platelet count >=70,000/ mm^3
* Blood chemistry results of:

  * albumin and direct bilirubin within normal limits
  * alpha fetoprotein (AFP) within reference range
  * AFP-L3<=10%
  * Protein induced by vitamin K (PIVKA)-II <=100 mAU/mL

Exclusion Criteria:

* Participants who did not previously respond virologically to combination therapy with interferon (including polyethylene glycol-modified interferon) and ribavirin
* Participants who had previously received treatment with interferon for whom at least 90 days have not elapsed since the end of previous treatment
* Participants who have received treatment within 14 days prior to registration with injectable preparations containing glycyrrhizin/cysteine/glycyron or shosaikoto
* Participants who have received administration of drugs having antiviral, anti-tumor, or immuno-modulating effect (including glucocorticoids and radiation therapy) within 90 days prior to registration (excluding local administration and topicals)
* Participants who have received other investigational drugs within 180 days prior to registration
* Hepatitis B surface (HBs) antigen positive
* Antinuclear antibody >=320 times
* Serum creatinine exceeding the upper limit of reference range
* Participants with fasting blood glucose >=110 mg/dL (participants with fasting blood glucose >=110 mg/dL and <126 mg/dL can be registered if their hemoglobin A1C (HbA1c) is <6.5%) [fasting blood glucose should be measured when participants are not receiving treatment for diabetes mellitus]
* Participants with any of the following: diabetes mellitus that requires treatment; thyroid function disorder not controlled by treatment; liver disease such as autoimmune, alcoholic and drug-induced liver diseases; hemophilia; arrhythmia requiring treatment; co-existing hypertension not controlled by drug therapy (systolic blood pressure [BP] >=160mmHg or diastolic BP>=100mmHg); chronic pulmonary disease; hemoglobinopathies (thalassemia, sickle cell anemia); malignant tumors or who have a history of malignant tumor within the past 5 years; organ transplants (other than cornea and hair transplant)
* Participants with or who have a history of primary biliary cirrhosis, liver failure, hepatic carcinoma; decompensated liver cirrhosis with any the following diseases: ascites, jaundice, variceal hemorrhage, esophageal or gastric varices requiring treatment, hepatic encephalopathy, and idiopathic bacterial peritonitis; depression or schizophrenia requiring treatment, or suicidal attempt or suicidal ideation; epileptic seizures requiring treatment; angina, cardiac failure, myocardial infarction, or life-threatening arrhythmia; autoimmune disease (Hashimoto's disease, Crohn's disease, ulcerative colitis, chronic rheumatoid arthritis, idiopathic thrombocytopenic purpura, systemic erythematosus, autoimmune hemolytic anemia, scleroderma, etc.); hepatic carcinoma
* Participants with a history of hypersensitivity to interferon preparations, biological products such as vaccine, or nucleoside analogs, and those with specific reaction to pegylated interferon alfa-2b in the prick test conducted before the initiation of treatment
* Women who are pregnant or nursing as well as women for whom pregnancy cannot be ruled out by serum human chorionic gonadotropin (HCG) test conducted during the screening period. Male participants with partners who are pregnant.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2007-06; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

IPD SHARING:
Plan to Share IPD: Yes
http://www.merck.com/clinical-trials/pdf/Merck%20Procedure%20on%20Clinical%20Trial%20Data%20Access%20Final_Updated%20July_9_2014.pdf
  http://engagezone.msd.com/ds_documentation.php

RESULTS

PARTICIPANT FLOW:
Groups:
- Peginterferon Alfa-2b + Ribavirin: Peginterferon alfa-2b administered at 1.0 µg/kg/week SC for 48 weeks plus ribavirin administered based on body weight and hemoglobin value at screening: 600-1000 mg/day
  for subjects with hemoglobin value at screening >=14g/dL, and 400-800 mg/day for subjects with hemoglobin value at screening >=12g/dL and <14g/dL for 48 weeks
Period: Overall Study
Arm/Group | Peginterferon Alfa-2b + Ribavirin
Started | 102
Completed | 51
Not Completed | 51
Not completed — Adverse Event | 8
Not completed — Discontinuance criteria met | 7
Not completed — HCV-RNA positive conversion | 34
Not completed — Withdrawal by Subject | 1
Not completed — Lack of Efficacy | 1

BASELINE CHARACTERISTICS:
Arm/Group | Peginterferon Alfa-2b + Ribavirin
Number analyzed (Participants) | 102
Age, Continuous [Mean (Standard Deviation); unit: Years] | 58.6 (8.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 48
  Male | 54
Region of Enrollment [Number; unit: Participants]
  Japan | 102

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Undetectable HCV-RNA at Week 72 (Sustained Virologic Response)
Description: Serum HCV-RNA was qualitatively measured by reverse transcriptase polymerase chain reaction (RT-PCR)
Time Frame: Measured at 24 weeks after 48 weeks treatment (72 weeks)
Measure: Number; unit: Participants
Arm/Group | Peginterferon Alfa-2b + Ribavirin
Number analyzed (Participants) | 102
Participants
  Undetectable HCV-RNA | 41
  Detectable HCV-RNA | 40
  Unknown (data not available) | 21

2. Secondary Outcome: Number of Participants With Undetectable HCV-RNA at Week 24
Description: Serum HCV-RNA was qualitatively measured by reverse transcriptase polymerase chain reaction (RT-PCR)
Time Frame: Week 24
Population: Peginterferon alfa-2b administered at 1.0 μg/kg/week SC for 48 weeks plus ribavirin administered based on body weight and hemoglobin value at screening: 600-1000 mg/day for subjects with hemoglobin value at screening >=14g/dL, and 400-800 mg/day for subjects with hemoglobin value at screening >=12g/dL and <14g/dL for 48 weeks
Measure: Number; unit: Participants
Arm/Group | Peginterferon Alfa-2b + Ribavirin
Number analyzed (Participants) | 102
Participants
  Undetectable HCV-RNA | 61
  Detectable HCV-RNA | 35
  Unknown (data not available) | 6

3. Secondary Outcome: Number of Participants With Undetectable HCV-RNA at End of Treatment
Description: Serum HCV-RNA was qualitatively measured by reverse transcriptase polymerase chain reaction (RT-PCR)
Time Frame: Up to 48 weeks
Measure: Number; unit: Participants
Arm/Group | Peginterferon Alfa-2b + Ribavirin
Number analyzed (Participants) | 102
Participants
  Undetectable HCV-RNA | 59
  Detectable HCV-RNA | 43
  Unknown (data not available) | 0

ADVERSE EVENTS:
Arm/Group | Peginterferon Alfa-2b + Ribavirin
Serious Adverse Events (participants affected / at risk) | 14/102
Other Adverse Events (participants affected / at risk) | 102/102
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Peginterferon Alfa-2b + Ribavirin (N=102)
ATRIAL FIBRILLATION (Cardiac disorders) | 1 (1)
CATARACT (Eye disorders) | 2 (2)
DIPLOPIA (Eye disorders) | 1 (1)
VARICES OESOPHAGEAL (Gastrointestinal disorders) | 1 (1)
MALAISE (General disorders) | 1 (1)
BURSITIS INFECTIVE (Infections and infestations) | 1 (1)
PNEUMONIA (Infections and infestations) | 1 (1)
SKIN LACERATION (Injury, poisoning and procedural complications) | 1 (1)
HEPATIC NEOPLASM MALIGNANT (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4)
LYMPHOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
CEREBRAL INFARCTION (Nervous system disorders) | 1 (1)
SUBARACHNOID HAEMORRHAGE (Nervous system disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Peginterferon Alfa-2b + Ribavirin (N=102)
PALPITATIONS (Cardiac disorders) | 6 (7)
EYE PRURITUS (Eye disorders) | 8 (8)
ABDOMINAL DISCOMFORT (Gastrointestinal disorders) | 17 (18)
ABDOMINAL PAIN (Gastrointestinal disorders) | 12 (14)
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 7 (8)
CONSTIPATION (Gastrointestinal disorders) | 18 (22)
DIARRHOEA (Gastrointestinal disorders) | 20 (28)
NAUSEA (Gastrointestinal disorders) | 37 (48)
STOMATITIS (Gastrointestinal disorders) | 25 (30)
VARICES OESOPHAGEAL (Gastrointestinal disorders) | 6 (6)
VOMITING (Gastrointestinal disorders) | 13 (17)
CHILLS (General disorders) | 6 (6)
INJECTION SITE ERYTHEMA (General disorders) | 43 (47)
INJECTION SITE PRURITUS (General disorders) | 27 (30)
INJECTION SITE RASH (General disorders) | 10 (11)
MALAISE (General disorders) | 90 (103)
OEDEMA PERIPHERAL (General disorders) | 8 (9)
PYREXIA (General disorders) | 96 (122)
THIRST (General disorders) | 11 (11)
HEPATIC STEATOSIS (Hepatobiliary disorders) | 6 (6)
NASOPHARYNGITIS (Infections and infestations) | 36 (54)
PHARYNGITIS (Infections and infestations) | 6 (7)
CONTUSION (Injury, poisoning and procedural complications) | 7 (7)
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 26 (28)
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 31 (32)
BASOPHIL COUNT INCREASED (Investigations) | 17 (20)
BILIRUBIN CONJUGATED INCREASED (Investigations) | 8 (10)
BLOOD ALBUMIN DECREASED (Investigations) | 7 (7)
BLOOD AMYLASE INCREASED (Investigations) | 33 (44)
BLOOD BILIRUBIN INCREASED (Investigations) | 18 (25)
BLOOD BILIRUBIN UNCONJUGATED INCREASED (Investigations) | 31 (36)
BLOOD CHLORIDE INCREASED (Investigations) | 9 (9)
BLOOD PHOSPHORUS DECREASED (Investigations) | 23 (25)
BLOOD POTASSIUM DECREASED (Investigations) | 15 (17)
BLOOD PRESSURE INCREASED (Investigations) | 9 (9)
BLOOD THYROID STIMULATING HORMONE DECREASED (Investigations) | 9 (9)
BLOOD THYROID STIMULATING HORMONE INCREASED (Investigations) | 18 (22)
BLOOD TRIGLYCERIDES INCREASED (Investigations) | 32 (39)
BLOOD URIC ACID INCREASED (Investigations) | 15 (16)
C-REACTIVE PROTEIN INCREASED (Investigations) | 11 (11)
EOSINOPHIL COUNT INCREASED (Investigations) | 19 (22)
GAMMA-GLUTAMYLTRANSFERASE INCREASED (Investigations) | 27 (28)
GLYCOSYLATED HAEMOGLOBIN DECREASED (Investigations) | 8 (9)
HAEMATOCRIT DECREASED (Investigations) | 82 (87)
HAEMOGLOBIN DECREASED (Investigations) | 91 (94)
HYALURONIC ACID INCREASED (Investigations) | 52 (59)
LIPASE INCREASED (Investigations) | 33 (45)
LYMPHOCYTE COUNT DECREASED (Investigations) | 89 (107)
LYMPHOCYTE COUNT INCREASED (Investigations) | 32 (45)
NEUTROPHIL COUNT DECREASED (Investigations) | 87 (113)
NEUTROPHIL COUNT INCREASED (Investigations) | 17 (21)
PLATELET COUNT DECREASED (Investigations) | 65 (76)
PROTEIN INDUCED BY VITAMIN K ABSENCE OR ANTAGONIST II INCREASED (Investigations) | 9 (9)
RED BLOOD CELL COUNT DECREASED (Investigations) | 86 (88)
RETICULOCYTE COUNT DECREASED (Investigations) | 6 (6)
RETICULOCYTE COUNT INCREASED (Investigations) | 8 (8)
RETICULOCYTE PERCENTAGE DECREASED (Investigations) | 15 (17)
RETICULOCYTE PERCENTAGE INCREASED (Investigations) | 56 (62)
THYROXINE FREE DECREASED (Investigations) | 8 (8)
TRI-IODOTHYRONINE FREE DECREASED (Investigations) | 9 (9)
WEIGHT DECREASED (Investigations) | 36 (36)
WHITE BLOOD CELL COUNT DECREASED (Investigations) | 94 (108)
DECREASED APPETITE (Metabolism and nutrition disorders) | 61 (77)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 56 (70)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 33 (36)
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 10 (11)
MUSCULOSKELETAL STIFFNESS (Musculoskeletal and connective tissue disorders) | 7 (10)
MYALGIA (Musculoskeletal and connective tissue disorders) | 56 (70)
DIZZINESS (Nervous system disorders) | 21 (24)
DIZZINESS POSTURAL (Nervous system disorders) | 9 (9)
DYSGEUSIA (Nervous system disorders) | 13 (14)
HEADACHE (Nervous system disorders) | 83 (111)
INSOMNIA (Psychiatric disorders) | 45 (52)
MOOD ALTERED (Psychiatric disorders) | 8 (8)
COUGH (Respiratory, thoracic and mediastinal disorders) | 21 (27)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 10 (10)
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 13 (16)
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 14 (14)
ALOPECIA (Skin and subcutaneous tissue disorders) | 47 (47)
DERMATITIS CONTACT (Skin and subcutaneous tissue disorders) | 6 (6)
DRY SKIN (Skin and subcutaneous tissue disorders) | 9 (9)
ECZEMA (Skin and subcutaneous tissue disorders) | 10 (11)
ERYTHEMA (Skin and subcutaneous tissue disorders) | 12 (12)
PRURITUS (Skin and subcutaneous tissue disorders) | 34 (42)
PRURITUS GENERALISED (Skin and subcutaneous tissue disorders) | 9 (10)
RASH (Skin and subcutaneous tissue disorders) | 40 (47)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No